CLINICAL TRIAL: NCT02513433
Title: Comparative Evaluation of Newer Congeners i.e. Levobupivacaine and Ropivacaine With Bupivacaine, in Lumbar Epidural Anaesthesia for Hip Surgeries
Brief Title: Comparison of Levobupivacaine, Ropivacaine and Bupivacaine in Epidural Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Government Medical College, Haldwani (Other)
Responsible Party: Principal Investigator, Dr Subhro Mitra, Assistant Professor, Government Medical College, Haldwani
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 65/IEC/01/12-13
Record Dates: First submitted 2015-07-30; First posted 2015-07-31 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-07

CONDITIONS: Pain Insensitivity, Congenital
Keywords: Lumbar epidural anaesthesia
MeSH Terms: conditions — Pain Insensitivity, Congenital | interventions — Bupivacaine; Levobupivacaine; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bupivacaine & Levobupivacaine (Active Comparator): Bupivacaine 15 ml 0.5% and Levobupivacaine 15 ml 0.5% in epidural route before surgery
  Interventions: Drug: Bupivacaine; Drug: Levobupivacaine
- Bupivacaine & Ropivacaine (Active Comparator): Bupivacaine 15 ml 0.5% and Ropivacaine 15 ml 0.75% in epidural route before surgery
  Interventions: Drug: Bupivacaine; Drug: Ropivacaine
- Ropivacaine & Levobupivacaine (Active Comparator): Ropivacaine 15 ml 0.75% and Levobupivacaine 15 ml 0.5% in epidural route before surgery
  Interventions: Drug: Levobupivacaine; Drug: Ropivacaine

INTERVENTIONS:
Drug: Bupivacaine — Local anesthetic
  Other Names: Anawin; Sensorcaine
  Arms: Bupivacaine & Levobupivacaine; Bupivacaine & Ropivacaine
Drug: Levobupivacaine — Local anesthetic
  Other Names: Levo-anawin
  Arms: Bupivacaine & Levobupivacaine; Ropivacaine & Levobupivacaine
Drug: Ropivacaine — Local anesthetic
  Other Names: Ropin
  Arms: Bupivacaine & Ropivacaine; Ropivacaine & Levobupivacaine

SUMMARY:
This study compares the clinical efficacy of newer local anaesthetic drugs Levobupivacaine and Ropivacaine with Bupivacaine in lumbar epidural anaesthesia for hip surgeries.

DETAILED DESCRIPTION:
Some of the most common day care surgeries are hip surgeries, in which local anaesthetic agents can be used via epidural route for both intra-op and post-op analgesia.

Among the drugs used nowadays are Lignocaine, Bupivacaine, Levobupivacaine and Ropivacaine.However Bupivacaine usage is not free from side effects.

The claimed benefits of both Levobupivacaine and Ropivacaine are reduced cardiac toxicity on overdose and more specific effects on sensory rather than motor nerve fibres.

Ropivacaine, an analog of Mepivacaine, is one of the long acting amide anaesthetic agent similar to Bupivacaine in chemical structure and anaesthetic function. It is a first enantiomer-specific compound, which has a reduced risk of cardio toxicity, neuro toxicity and rapid recovery of motor function. Levobupivacaine is the pure S (-)-enantiomer of Bupivacaine, and in recent year has emerged as a safer alternative for regional anaesthesia than its racemic parent.

ELIGIBILITY:
Inclusion Criteria:

* ASA Grade I and II patients of either sex
* Age 18-60 years
* Undergoing various hip surgeries under lumbar epidural anesthesia

Exclusion Criteria:

* Refusal for epidural
* ASA-III&IV
* Head injury
* Psychiatric disease
* Known allergic to test drugs
* Major systemic disease
* Any analgesia with in past 24 hours

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2012-12; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Onset of sensory block | 30 minutes
  Time to achieve sensory block up to tenth thoracic dermatome

SECONDARY OUTCOMES:
Time for 2 segment regression of sensory block | 90 minutes
  Time for regression of sensory block 2 segments lower than maximum blocked dermatome
Time to achieve maximum motor block | 45 minutes
  Time to achieve motor block of modified Bromage score

CONTACTS AND LOCATIONS:
Overall Officials: Geeta Bhandari, M.D., Principal Investigator — Professor and Head of the department
Locations (1):
- Government Medical College, Haldwani, Uttarakhand, India